CLINICAL TRIAL: NCT06584903
Title: Fan Use During Extreme Heat: Safe Thermal Limits
Brief Title: Safe Indoor Temperature Limit for Fans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Nicholas Ravanelli, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 26897
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heat Exposure; Healthy; Young Adults; Fans
Keywords: indoor temperature; core temperature; heart rate; electric fans; cardiovascular strain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Still air (Placebo Comparator): still air condition with no supplemental air flow
  Interventions: Other: Temperature Ramp Protocol
- Electric fan (Experimental): Force air flow with a 46 cm 3-blade fan positioned 1.2 m anterior to the participants chest
  Interventions: Other: Temperature Ramp Protocol

INTERVENTIONS:
Other: Temperature Ramp Protocol — Following a 45 minute baseline in 37°C seated on a chair, the indoor temperature in the climate-controlled room increased from 37°C to 47°C at ~0.06°C/min (relative humidity ~26%) over 180 minutes.

SUMMARY:
Extreme heat events are a significant global threat to health and wellbeing, and result in more morbidity and mortality than all other natural disasters combined. Thus, a key priority is identifying effective and accessible heat resilience solutions to protect individuals from the potentially fatal consequences of heat stress. Within a range of ambient conditions, a fan has been recognized a low-cost heat resilience solution. However, when ambient temperatures exceed skin temperatures (e.g., above 35°C), a fan will incur greater dry heat gain which may be counterbalanced with evaporation of sweat from the skin surface. However, at a critical indoor temperature, the rate of heat gain will exceed the rate of evaporation resulting in net heat gain. The critical indoor temperature has yet to be determined. The purpose of this present study is to identify the indoor temperature at which a fan results in greater cardiovascular and thermal strain relative to still air in young adults using a simulated heat wave scenario of a warming room.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index less than 30
* male or female
* ability to tolerate hot environments for a prolonged period (e.g. >2 h)

Exclusion Criteria:

* Any respiratory disease
* Any cardiovascular disease, including hypertension
* Diabetes
* not currently on any medication (except oral contraceptives)

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | At baseline (e.g. 0 minutes), and every 10 minutes of exposure up to 180 minutes
  Measured with an electrocardiogram-gated automated cuff
Rate Pressure Product | At baseline (e.g. 0 minutes), and every 10 minutes of exposure up to 180 minutes
Heart Rate | At baseline (e.g. 0 minutes), and every minute for the 180 minute experimental trial
  Measured with a 3-lead electrocardiogram
Skin Temperature | At baseline (e.g. 0 minutes), and every minute for the 180 minute experimental trial
  Measured at 4 skin locations (chest, arm, thigh, and calf) using wireless iButtons affixed to the skin with surgical tape
Core Temperature | At baseline (e.g. 0 minutes), and every minute for the 180 minute experimental trial
  rectal temperature measured with a pediatric grade thermistor probe
Whole-Body Sweat Rate | At baseline (e.g. 0 minutes), and every minute for the 180 minute experimental trial
  Net difference in body mass (pre versus post) using a balance scale placed below the chair of the participant

SECONDARY OUTCOMES:
Thermal Sensation | At baseline (e.g. 0 minutes), and every 10 minutes for the 180 minute experimental trial
  visual analog scale
Thermal comfort | Assessed at baseline (e.g. 0 minutes), and every 10 minutes for the 180 minute experimental trial
  visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ravanelli, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All deidentified participant data supporting the findings of this study will be made freely available on the Open Science Framework Repository.
Time Frame: Following publication
Access Criteria: Anyone will be allowed to access the data supporting the findings through the Open Science Framework Repository.